CLINICAL TRIAL: NCT01361022
Title: A Randomized, Single-dose, Two-way Cross-over Study to Assess the Bioequivalence of Lendormin Tablets 0.25 mg (Delpharm Reims) vs. Lendormin Tablets 0.25 mg (Synmosa Biopharma Co. Ltd.) Administered to Healthy Adult Volunteers
Brief Title: To Assess the Bioequivalence of Brotizolam Tablets 250 Mcg vs. Lendormin Tablets 250 Mcg Administered to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 263.511
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — brotizolam

ARMS (2):
- Brotizolam tablet (Active Comparator): Brotizolam tablets 250mcg : at least 6 and 24 subjects will be enrolled in the pre-study and main study, respectively
  Interventions: Drug: Brotizolam tablet
- Lendormin tablet (Experimental): Lendormin tablets 250mcg: at least 6 and 24 subjects will be enrolled in the pre-study and main study, respectively
  Interventions: Drug: Lendormin tablet

INTERVENTIONS:
Drug: Lendormin tablet — Lendormin tablet 250mc is administrated and compared
  Arms: Lendormin tablet
Drug: Brotizolam tablet — Brotizolam tablet 250mc is administrated and compared
  Arms: Brotizolam tablet

SUMMARY:
The objective of the study was to assess the bioequivalence of Lendormin Tablets (Delpharm Reims) vs. Lendormin Tablets (Synmosa Biopharma Co. Ltd.) following oral administration

ELIGIBILITY:
Inclusion criteria:

1. Healthy volunteers, provision of signed written informed consent before enrolment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
2. Healthy adult male, aged between 20 and 40 years old.
3. Body Mass Index (BMI) between 18.5 and 25, inclusive, (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2]).
4. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest x-ray and electrocardiogram.
5. No significant deviation from normal biochemistry examination.
6. No significant deviation from normal haematology examination.
7. No significant deviation from normal urinalysis examination.

Exclusion criteria:

1. History of drug or alcohol abuse within the past one year.
2. Medical history of allergic asthma or sensitivity to analogous drug.
3. Evidence of chronic or acute infectious diseases from 4 weeks before the study.
4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology.
5. Ongoing peptic ulcer and constipation.
6. Planned vaccination during the time course of the study.
7. Taking any clinical investigation drug from 3 months before the study.
8. Use of any medication, including herb medicine or vitamins from 4 weeks before the study.
9. Donation of greater than 250 ml of blood in the past 3 months prior to dosing or donation of 250 ml of blood in the past 2 months prior to dosing.
10. A positive Hepatitis B surface antigen or positive Hepatitis C antibody result.
11. A positive test for HIV(Human immunodeficiency virus) antibody.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Cmax: Peak drug concentration obtained directly from the data without interpolation | One month
kel:Plasma elimination rate constant determined by simple linear regression based on the terminal phase of plasma concentration | One month
Tmax:Time to peak drug concentration obtained directly from the data without interpolation | One month
T 1/2: Plasma half-life estimated by (0.693/kel) | One month
MRT : Mean residence time | One month
AUMC : Area under the ( first) moment plasma concentration - time curve | One month
AUC 0-t: Area under the plasma concentration-time curve from zero to the last quantifiable concentration determined by the traperoidal rule | One month
AUC 0- : Area under the plasma concentration-time curve from time zero to infinity determined by the trapezoidal rule and extrapolated to infinity estimated by the last quantifiable concentration (Cn) divided by kel | One month

SECONDARY OUTCOMES:
Blood pressure | one month
heart rate | one month
body temperature | One month
12 Laed ECG, Lab Test ( Hematocrit, WBC count with differential, RBC count and platelet count ; SGOT ( AST), SGPT (ALT) , alkaline phosphatase, total bilirubin, albumin, glucose, BUN, creatinine,uric acid, total cholesterol and TG) | One month

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 263.511.1 Boehringer Ingelheim Investigational Site, Taipei, Taiwan